CLINICAL TRIAL: NCT04110925
Title: Mutational Analysis as a Prognostic and Predictive Marker of Cardiovascular Disease in Patients With Myelodysplasia
Brief Title: Mutational Analysis as a Prognostic and Predictive Marker of Cardiovascular (CVD) Disease in Patients With Myelodysplasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Ontario Molecular Pathology Research Network (Unknown); Queen's University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: MDS CVD
Record Dates: First submitted 2019-08-23; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: MDS; Cardiovascular Diseases; Inflammation
Keywords: CT imaging; next generation sequencing; myelodysplastic syndrome
MeSH Terms: conditions — Cardiovascular Diseases; Inflammation; Myelodysplastic Syndromes | interventions — Mutation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MDS patients (Other): All Canadian MDS patients on the MDS-database to be included.
  Interventions: Genetic: Genetic Mutations; Other: Inflammatory and lipid markers; Other: Computed Tomography (CT) of the heart

INTERVENTIONS:
Genetic: Genetic Mutations — DNA sequencing for mutations to be obtained by bloodwork within 6 months of diagnosis, or by accessing diagnostic bone marrow aspirate slides.
Other: Inflammatory and lipid markers — Bloodwork to be done for lipid profile, c-reactive protein (CRP), and multiplex chemokine/cytokine analysis.
Other: Computed Tomography (CT) of the heart — Sunnybrook Patients with no history of cardiovascular disease [ex: past/present coronary artery disease (CAD), peripheral vascular disease (PVD), angina, myocardial infarction (MI), stroke, transient ischemic attack (TIA), or stents], not pregnant, and able to undergo CT will receive a CT of the heart to look for and quantify any occult coronary artery disease.

SUMMARY:
This study evaluates the relationship between myelodysplastic syndromes (MDS) and cardiovascular disease. MDS patients will be evaluated for the presence of mutations and whether they are associated with an increased risk of heart disease (CVD) and inflammation compared to healthy adults. Patients without symptoms of CVD will receive CT scans to assess for hidden disease and if that is related to their mutations.

DETAILED DESCRIPTION:
Myelodysplastic syndromes (MDS) are a type of blood cancer that can cause infection or bleeding because they prevent the formation of blood components and may lead to leukemia and death. MDS can arise from changes (or mutations) to a patient's DNA. MDS patients have increased risk of heart disease compared to healthy adults. The investigators will look for links between mutations in MDS patients and increased risk of heart disease. They will also use "CT imaging" to see if MDS patients have asymptomatic artery disease but may lead to heart disease in the future and if that is related to their mutations. The researcher will try to link mutations in MDS patients to markers of inflammation and to the amount of artery disease on CT imaging to look for patterns. The goal is to find certain mutations that are associated with inflammation and heart disease. This may ultimately allow hematologists to test MDS patients with these mutations for heart disease and/or treat them early so they have a better and longer life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of: myelodysplastic syndrome (MDS), myeloproliferative neoplasm (MPN), Chronic myelomonocytic leukemia leukemia (CMML), or low-blast acute myeloid leukemia (AML, blasts 20-29%) less than 24 months ago
* Alive and registered in the MDS-Canada (MDS-CAN) database
* Known comorbidity history and known history of cardiovascular disease
* Able to provide peripheral blood sample for cytokine analysis
* Able top provide samples for next generation sequencing (NGS) - if diagnosis 0-6 months ago: peripheral blood; if diagnosis 6-24 months ago: diagnostic bone marrow aspirate slides or peripheral blood

Exclusion Criteria:

* MDS/MPN patients other than CMML due to higher prevalence of Janus Kinase 2 (JAK2) mutation (a known risk factor for CVD)
* Disease progression without available diagnostic bone marrow slides for NGS

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Measure the allelic frequency and type of myeloid cancer-associated mutations in MDS patients diagnostic bone marrow aspirates or slides | 2 years
  Screen for Presence of myeloid-cancer associated mutations and their variant allele frequencies (VAF) at diagnosis of MDS as measured through next generation sequencing of 40 myeloid genes.
Screen for occult and potentially clinically significant CAD in MDS patients by means of coronary CT | 2 years
  Patients at Sunnybrook hospital with no pre-existing history of CAD who receive CT of the heart and found to harbour occult CAD by means of coronary calcium scoring:
  1. zero calcium (No CAD)
  2. 1-400: mild-moderate calcification
  3. >400: severe calcification
Identify any correlation between selected myeloid mutations and/or their VAF with the presence of pre-existing incident or occult CAD | 2 years
  Comparing the presence of myeloid-cancer associated mutations and their variant allele frequencies (VAF) at diagnosis of MDS as measured through next generation sequencing of 40 myeloid genes between patients with pre-existing/occult CAD and those without.

SECONDARY OUTCOMES:
Track how often newly discovered CAD from coronary CT leads to further intervention or changes in monitoring | 2 years
  The investigators will track any interventions in patients without a prior history of CAD who who are discovered to have occult CAD by coronary CT. This includes number of patients who were recommended:
  1. medical management of CAD
  2. Referral to clinical cardiologist
  3. Invasive angiography
Screen for serum inflammatory cytokines in the blood of patients with incident or occult CAD | 2 years
  Measure TNFa, IL-1beta, IL-6 and an array of other inflammatory cytokines (to be determined) in the peripheral blood upon enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Rashmi S Goswani, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Stahl M, Zeidan AM. Management of lower-risk myelodysplastic syndromes without del5q: current approach and future trends. Expert Rev Hematol. 2017 Apr;10(4):345-364. doi: 10.1080/17474086.2017.1297704. Epub 2017 Mar 9. PMID 28277851
- [Background] Brunner AM, Blonquist TM, Hobbs GS, Amrein PC, Neuberg DS, Steensma DP, Abel GA, Fathi AT. Risk and timing of cardiovascular death among patients with myelodysplastic syndromes. Blood Adv. 2017 Oct 18;1(23):2032-2040. doi: 10.1182/bloodadvances.2017010165. eCollection 2017 Oct 24. PMID 29296849
- [Background] Papaemmanuil E, Gerstung M, Malcovati L, Tauro S, Gundem G, Van Loo P, Yoon CJ, Ellis P, Wedge DC, Pellagatti A, Shlien A, Groves MJ, Forbes SA, Raine K, Hinton J, Mudie LJ, McLaren S, Hardy C, Latimer C, Della Porta MG, O'Meara S, Ambaglio I, Galli A, Butler AP, Walldin G, Teague JW, Quek L, Sternberg A, Gambacorti-Passerini C, Cross NC, Green AR, Boultwood J, Vyas P, Hellstrom-Lindberg E, Bowen D, Cazzola M, Stratton MR, Campbell PJ; Chronic Myeloid Disorders Working Group of the International Cancer Genome Consortium. Clinical and biological implications of driver mutations in myelodysplastic syndromes. Blood. 2013 Nov 21;122(22):3616-27; quiz 3699. doi: 10.1182/blood-2013-08-518886. Epub 2013 Sep 12. PMID 24030381
- [Background] Elbaek MV, Sorensen AL, Hasselbalch HC. Cardiovascular disease in chronic myelomonocytic leukemia: do monocytosis and chronic inflammation predispose to accelerated atherosclerosis? Ann Hematol. 2019 Jan;98(1):101-109. doi: 10.1007/s00277-018-3489-0. Epub 2018 Sep 4. PMID 30182347
- [Background] Jaiswal S, Natarajan P, Silver AJ, Gibson CJ, Bick AG, Shvartz E, McConkey M, Gupta N, Gabriel S, Ardissino D, Baber U, Mehran R, Fuster V, Danesh J, Frossard P, Saleheen D, Melander O, Sukhova GK, Neuberg D, Libby P, Kathiresan S, Ebert BL. Clonal Hematopoiesis and Risk of Atherosclerotic Cardiovascular Disease. N Engl J Med. 2017 Jul 13;377(2):111-121. doi: 10.1056/NEJMoa1701719. Epub 2017 Jun 21. PMID 28636844
- [Background] Okwuosa TM, Greenland P, Ning H, Liu K, Bild DE, Burke GL, Eng J, Lloyd-Jones DM. Distribution of coronary artery calcium scores by Framingham 10-year risk strata in the MESA (Multi-Ethnic Study of Atherosclerosis) potential implications for coronary risk assessment. J Am Coll Cardiol. 2011 May 3;57(18):1838-45. doi: 10.1016/j.jacc.2010.11.053. PMID 21527159